CLINICAL TRIAL: NCT00316888
Title: Phase II Trial of Cetuximab Plus Cisplatin, 5- Fluorouracil and Radiation in Immunocompetent Patients With Anal Carcinoma
Brief Title: Cetuximab, Cisplatin, Fluorouracil, and Radiation Therapy in Treating Patients With Anal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ECOG-ACRIN Cancer Research Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: Eastern Cooperative Oncology Group (Network)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E3205; E3205 (Other: ECOG-ACRIN Cancer Research Group); U10CA023318 (NIH); CDR0000470269 (Registry Identifier: Clinical Data Repository)
Record Dates: First submitted 2006-04-19; First posted 2006-04-21 (Estimated); Results first posted 2016-08-29 (Estimated); Last update posted 2023-06-29 (Actual); Status verified 2023-06

CONDITIONS: Anal Cancer
Keywords: squamous cell carcinoma of the anus; stage I anal cancer; stage II anal cancer; stage IIIA anal cancer; stage IIIB anal cancer; basaloid carcinoma of the anus; cloacogenic carcinoma of the anus
MeSH Terms: conditions — Anus Neoplasms; Anal Canal Carcinoma | interventions — Cetuximab; Cisplatin; Fluorouracil; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm I (closed to accrual as of 11/3/2008) (Experimental): Patients receive cisplatin IV over 60 minutes on days 1, 29, 57, and 85 and fluorouracil IV continuously over 96 hours on days 1-4, 29-32, 57-60, and 85-88. Patients also receive cetuximab IV over 120 minutes on day 50 and then IV over 60 minutes on days 57, 64, 71, 78, 85, 92, and 99 and undergo radiotherapy once daily 5 days a week for 5 weeks, beginning on day 57. Treatment continues in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: cetuximab; Drug: cisplatin; Drug: fluorouracil; Radiation: radiotherapy
- Arm II (open to accrual on 8/18/2009) (Experimental): Patients receive cetuximab IV over 120 minutes on day 1 and then IV over 60 minutes on days 8, 15, 22, 29, 36, 43, and 50. Patients also receive cisplatin IV over 60 minutes on days 1 and 36, fluorouracil IV continuously over 96 hours on days 8-11 and 36-39, and undergo radiotherapy once daily 5 days a week for 5 weeks beginning on day 8. Treatment continues in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: cetuximab; Drug: cisplatin; Drug: fluorouracil; Radiation: radiotherapy

INTERVENTIONS:
Biological: cetuximab — Given IV
  Other Names: Erbitux
Drug: cisplatin — Given IV
  Other Names: Cis-diaminedichloroplatinum Cis-diaminedichloroplatinum (II); Platinol; Platinol-AQ; cis-platinum; diaminedichloroplatinum; DDP
Drug: fluorouracil — Given IV
  Other Names: 5-Fluorouracil; 5-FU; Adrucil; Efudex
Radiation: radiotherapy — Given once daily 5 days a week for 5 weeks
  Other Names: radiation therapy

SUMMARY:
RATIONALE: Monoclonal antibodies, such as cetuximab, can block tumor growth in different ways. Some find tumor cells and kill them or carry tumor-killing substances to them. Others interfere with the ability of tumor cells to grow and spread. Drugs used in chemotherapy, such as cisplatin and fluorouracil, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Radiation therapy uses high-energy x-rays to kill tumor cells. Cetuximab may help cisplatin and fluorouracil work better by making tumor cells more sensitive to the drugs. It may also make tumor cells more sensitive to radiation therapy. Giving cetuximab together with chemotherapy and radiation therapy may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving cetuximab together with cisplatin, fluorouracil, and radiation therapy works in treating immunocompetent patients with stage I (closed to accrual as of 11/3/2008), stage II, (some stage II closed to accrual as of 11/3/2008) or stage III anal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary Objective:

* Determine whether the addition of cetuximab to combined modality therapy (CMT) comprising cisplatin, fluorouracil, and radiotherapy reduces the local failure rate by ≥ 50% at 3 years (compared with historical data) in immunocompetent patients with stage I-III invasive anal carcinoma.

Secondary Objectives:

* Determine objective response rate (complete and partial), progression-free survival, colostomy-free survival, and overall survival.
* Determine the overall toxicity of concurrent cisplatin, fluorouracil, and radiation therapy combined with cetuximab.

Exploratory Objectives:

* Evaluate the effect of cetuximab and CMT on anogenital herpes papilloma virus (HPV) infection and anal cytology.
* Evaluate whether moderate to strong expression of epidermal growth factor receptor, Phosphatidylinositol-4,5-bisphosphate 3-kinase (PI3K), and P-Akt (as determined by immunohistochemistry) is associated with an increased risk of local failure.

OUTLINE: This is a multicenter study with two sequential arms. Arm I was closed to accrual as of 11/3/2008, and arm II opened to accrual on 8/18/2009. Patients are assigned to 1 of the 2 treatment arms.

* Arm I (closed to accrual as of 11/3/2008): Patients receive cisplatin intravenously (IV) over 60 minutes on days 1, 29, 57, and 85 and fluorouracil IV continuously over 96 hours on days 1-4, 29-32, 57-60, and 85-88. Patients also receive cetuximab IV over 120 minutes on day 50 and then IV over 60 minutes on days 57, 64, 71, 78, 85, 92, and 99 and undergo radiotherapy once daily 5 days a week for 5 weeks, beginning on day 57.
* Arm II (open to accrual on 8/18/2009): Patients receive cetuximab IV over 120 minutes on day 1 and then IV over 60 minutes on days 8, 15, 22, 29, 36, 43, and 50. Patients also receive cisplatin IV over 60 minutes on days 8 and 36, fluorouracil IV continuously over 96 hours on days 8-11 and 36-39, and undergo radiotherapy once daily 5 days a week for 5 weeks beginning on day 8.

After completion of study treatment, patients are followed periodically for up to 10 years.

PROJECTED ACCRUAL: A total of 62 patients will be accrued for this study.

ELIGIBILITY:
INCLUSION CRITERIA:

* Histologically confirmed anal canal or perianal (anal margin) squamous cell carcinoma

  * Stage I-IIIB (closed to accrual as of 11/3/2008)
  * Stage II (T3, N0 only), IIIA, or IIIB
  * Tumors of nonkeratinizing histology, such as basaloid, transitional cell, or cloacogenic histology, allowed
  * No well-differentiated stage I anal margin cancer
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Hemoglobin ≥ 10 g/dL
* Platelet count ≥ 100,000/mm^3
* Absolute neutrophil count > 1,500/mm^3
* Creatinine ≤ 1.5 times upper limit of normal (ULN) OR creatinine clearance > 60 mL/min
* Bilirubin ≤ 2 times ULN
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) < 3 times ULN
* Negative pregnancy test
* Fertile patients must use effective contraception during and for ≥ 3 months after completion of study treatment
* No other malignancies except nonmelanomatous skin cancer

  * Prior malignancies must be in remission for ≥ 5 years
* Patients with a known risk factor for human immunodeficiency virus (HIV) infection must undergo HIV testing within 90 days before study entry AND must be HIV negative by antibody detection, culture, or quantitative assay of plasma HIV ribonucleic acid (RNA)

EXCLUSION CRITERIA:

* Presence of the following conditions within the past 6 months:

  * Active infection
  * Uncontrolled diabetes
  * New York Heart Association class II-IV congestive heart failure
  * Cerebrovascular accident
  * Transient ischemic attack
  * Uncontrolled hypertension
  * Unstable angina
  * Myocardial infarction
* History of rheumatic disorders, irritable bowel syndrome, or inflammatory bowel disease
* Known HIV positivity
* Known risk factors for HIV infection
* Prior radiotherapy or chemotherapy for this malignancy
* Prior pelvic radiotherapy
* Prior potentially curative surgery (i.e., abdominal or peritoneal resection) for anal cancer
* Pregnant or nursing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2007-02-28 (Actual); Primary Completion 2015-11 (Actual); Study Completion 2021-08-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Madhur K. Garg, MD, Study Chair — Montefiore Medical Center; Joseph A. Sparano, MD, Study Chair — Montefiore Medical Center
Locations (125):
- United States (125):
  - Stanford Cancer Center, Stanford, California
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Front Range Cancer Specialists, Fort Collins, Colorado
  - Robert H. Lurie Comprehensive Cancer Center at Northwestern University, Chicago, Illinois
  - Hematology and Oncology Associates, Chicago, Illinois
  - Decatur Memorial Hospital Cancer Care Institute, Decatur, Illinois
  - Kellogg Cancer Care Center, Highland Park, Illinois
  - Provena St. Mary's Regional Cancer Center - Kankakee, Kankakee, Illinois
  - North Shore Oncology and Hematology Associates, Limited - Libertyville, Libertyville, Illinois
  - Cancer Care and Hematology Specialists of Chicagoland - Niles, Niles, Illinois
  - Swedish-American Regional Cancer Center, Rockford, Illinois
  - Hematology Oncology Associates - Skokie, Skokie, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - Indiana University Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - William N. Wishard Memorial Hospital, Indianapolis, Indiana
  - Cedar Rapids Oncology Associates, Cedar Rapids, Iowa
  - Mercy Regional Cancer Center at Mercy Medical Center, Cedar Rapids, Iowa
  - Siouxland Hematology-Oncology Associates, LLP, Sioux City, Iowa
  - Mercy Medical Center - Sioux City, Sioux City, Iowa
  - St. Luke's Regional Medical Center, Sioux City, Iowa
  - Cancer Center of Kansas, PA - Chanute, Chanute, Kansas
  - Cancer Center of Kansas, PA - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas, PA - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Cancer Center of Kansas, PA - Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Cancer Center of Kansas, PA - Liberal, Liberal, Kansas
  - Cancer Center of Kansas, PA - Newton, Newton, Kansas
  - Cancer Center of Kansas, PA - Parsons, Parsons, Kansas
  - Cancer Center of Kansas, PA - Pratt, Pratt, Kansas
  - Cancer Center of Kansas, PA - Salina, Salina, Kansas
  - Cancer Center of Kansas, PA - Wellington, Wellington, Kansas
  - Associates in Womens Health, PA - North Review, Wichita, Kansas
  - Cancer Center of Kansas, PA - Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas, PA - Wichita, Wichita, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Via Christi Cancer Center at Via Christi Regional Medical Center, Wichita, Kansas
  - Cancer Center of Kansas, PA - Winfield, Winfield, Kansas
  - Mary Bird Perkins Cancer Center - Baton Rouge, Baton Rouge, Louisiana
  - MBCCOP - LSU Health Sciences Center, New Orleans, Louisiana
  - Medical Center of Louisiana - New Orleans, New Orleans, Louisiana
  - Greater Baltimore Medical Center Cancer Center, Baltimore, Maryland
  - Hickman Cancer Center at Bixby Medical Center, Adrian, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - Community Cancer Center of Monroe, Monroe, Michigan
  - Mercy Memorial Hospital - Monroe, Monroe, Michigan
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy and Unity Cancer Center at Mercy Hospital, Coon Rapids, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Mercy and Unity Cancer Center at Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - HealthEast Cancer Care at St. John's Hospital, Maplewood, Minnesota
  - Minnesota Oncology - Maplewood, Maplewood, Minnesota
  - Virginia Piper Cancer Institute at Abbott - Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center - Minneapolis, Minneapolis, Minnesota
  - Humphrey Cancer Center at North Memorial Outpatient Center, Robbinsdale, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Park Nicollet Cancer Center, Saint Louis Park, Minnesota
  - Regions Hospital Cancer Care Center, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - St. Francis Cancer Center at St. Francis Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Willmar Cancer Center at Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology - Woodbury, Woodbury, Minnesota
  - Cancer Resource Center - Lincoln, Lincoln, Nebraska
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Immanuel Medical Center, Omaha, Nebraska
  - Alegant Health Cancer Center at Bergan Mercy Medical Center, Omaha, Nebraska
  - Lakeside Hospital, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - Carol G. Simon Cancer Center at Morristown Memorial Hospital, Morristown, New Jersey
  - Overlook Hospital, Summit, New Jersey
  - NYU Cancer Institute at New York University Medical Center, New York, New York
  - Albert Einstein Cancer Center at Albert Einstein College of Medicine, The Bronx, New York
  - Wood County Oncology Center, Bowling Green, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Riverside Methodist Hospital Cancer Care, Columbus, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Grant Medical Center Cancer Care, Columbus, Ohio
  - Mount Carmel Health - West Hospital, Columbus, Ohio
  - Doctors Hospital at Ohio Health, Columbus, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Community Cancer Center, Elyria, Ohio
  - Hematology Oncology Center, Elyria, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - Lima Memorial Hospital, Lima, Ohio
  - Strecker Cancer Center at Marietta Memorial Hospital, Marietta, Ohio
  - Northwest Ohio Oncology Center, Maumee, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Licking Memorial Cancer Care Program at Licking Memorial Hospital, Newark, Ohio
  - St. Charles Mercy Hospital, Oregon, Ohio
  - Toledo Clinic - Oregon, Oregon, Ohio
  - Southern Ohio Medical Center Cancer Center, Portsmouth, Ohio
  - Community Hospital of Springfield and Clark County, Springfield, Ohio
  - Flower Hospital Cancer Center, Sylvania, Ohio
  - Mercy Hospital of Tiffin, Tiffin, Ohio
  - Toledo Hospital, Toledo, Ohio
  - St. Vincent Mercy Medical Center, Toledo, Ohio
  - Medical University of Ohio Cancer Center, Toledo, Ohio
  - CCOP - Toledo Community Hospital, Toledo, Ohio
  - St. Anne Mercy Hospital, Toledo, Ohio
  - Toledo Clinic, Incorporated - Main Clinic, Toledo, Ohio
  - Fulton County Health Center, Wauseon, Ohio
  - Genesis - Good Samaritan Hospital, Zanesville, Ohio
  - Joan Karnell Cancer Center at Pennsylvania Hospital, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center - Philadelphia, Philadelphia, Pennsylvania
  - Hematology and Oncology Associates of Northeastern Pennsylvania, Scranton, Pennsylvania
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Fredericksburg Oncology, Incorporated, Fredericksburg, Virginia
  - Marshfield Clinic - Chippewa Center, Chippewa Falls, Wisconsin
  - Marshfield Clinic Cancer Care at Regional Cancer Center, Eau Claire, Wisconsin
  - UW Cancer Center Johnson Creek, Johnson Creek, Wisconsin
  - University of Wisconsin Paul P. Carbone Comprehensive Cancer Center, Madison, Wisconsin
  - Marshfield Clinic - Marshfield Center, Marshfield, Wisconsin
  - Marshfield Clinic - Lakeland Center, Minocqua, Wisconsin
  - Ministry Medical Group at Saint Mary's Hospital, Rhinelander, Wisconsin
  - Marshfield Clinic - Indianhead Center, Rice Lake, Wisconsin
  - Marshfield Clinic at Saint Michael's Hospital, Stevens Point, Wisconsin
  - Marshfield Clinic - Wausau Center, Wausau, Wisconsin
  - Marshfield Clinic - Weston Center, Weston, Wisconsin
  - Marshfield Clinic - Wisconsin Rapids Center, Wisconsin Rapids, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data may be made available upon request as per the ECOG-ACRIN Data Sharing Policy.

REFERENCES:
- [Background] Garg M, Lee JY, Kachnic LA, et al.: Phase II trials of cetuximab (CX) plus cisplatin (CDDP), 5-fluorouracil (5-FU) and radiation (RT) in immunocompetent (ECOG 3205) and HIV-positive (AMC045) patients with squamous cell carcinoma of the anal canal (SCAC): safety and preliminary efficacy results. [Abstract] J Clin Oncol 30 (Suppl 15): A-4030, 2012.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was activated on January 19, 2007 and accrued its first patient on February 28, 2007, 28 patients were enrolled to arm I (closed to accrual on 11/3/2008) and 35 patients were enrolled to arm II (open to accrual on 8/18/2009).
Groups:
- Arm I (Closed to Accrual as of 11/3/2008): Patients receive cisplatin IV over 60 minutes on days 1, 29, 57, and 85 and fluorouracil IV continuously over 96 hours on days 1-4, 29-32, 57-60, and 85-88. Patients also receive cetuximab IV over 120 minutes on day 50 and then IV over 60 minutes on days 57, 64, 71, 78, 85, 92, and 99 and undergo radiotherapy once daily 5 days a week for 5 weeks, beginning on day 57. Treatment continues in the absence of disease progression or unacceptable toxicity.
  cetuximab: Given IV
  cisplatin: Given IV
  fluorouracil: Given IV
  radiation therapy: Given once daily 5 days a week for 5 weeks
- Arm II (Open to Accrual on 8/18/2009): Patients receive cetuximab IV over 120 minutes on day 1 and then IV over 60 minutes on days 8, 15, 22, 29, 36, 43, and 50. Patients also receive cisplatin IV over 60 minutes on days 1 and 36, fluorouracil IV continuously over 96 hours on days 8-11 and 36-39, and undergo radiotherapy once daily 5 days a week for 5 weeks beginning on day 8. Treatment continues in the absence of disease progression or unacceptable toxicity.
  cetuximab: Given IV
  cisplatin: Given IV
  fluorouracil: Given IV
  radiation therapy: Given once daily 5 days a week for 5 weeks
Period: Overall Study
Arm/Group | Arm I (Closed to Accrual as of 11/3/2008) | Arm II (Open to Accrual on 8/18/2009)
Started | 28 | 35
Eligible | 28 | 35
Treated | 28 (Received induction and/or chemo+radiation therapy) | 34
Started Induction Chemotherapy | 28 | 0 (Induction chemotherapy was removed for patients on this arm)
Started Chemo+Radiation+Cetuximab | 27 (One patient did not start chemo+radiation therapy after completing induction therapy) | 34
Completed | 22 | 27
Not Completed | 6 | 8
Not completed — Adverse Event | 4 | 5
Not completed — Withdrawal by Subject | 2 | 2
Not completed — Not start protocol therapy | 0 | 1

BASELINE CHARACTERISTICS:
Population: all eligible and treated patients
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Closed to Accrual as of 11/3/2008) | Arm II (Open to Accrual on 8/18/2009) | Total
Number analyzed (Participants) | 27 | 34 | 61
Age, Continuous [Median (Full Range); unit: years] | 56 [42 to 77] | 56 [37 to 78] | 56 [37 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 28 | 49
  Male | 6 | 6 | 12

OUTCOME MEASURES:

1. Primary Outcome: Local Failure Rate at 3 Years
Description: Local failure was defined as progression/relapse of disease in the anal canal and/or regional organs and/or regional lymph nodes after completion of protocol therapy, or progression during protocol therapy. Lost to follow-up and death (regardless of cause of death) prior to 3 years were also considered as local failures. For the calculation of local failure rate at 3 years, patients were classified into two groups (ie, coded as binary variable): failure (patients with local failure events prior to 3 years) vs. no failure (patients who still alive and had no local failure at 3 years). The binomial proportion and its exact two-sided 80% confidence interval (CI) were used to estimate it.
Time Frame: assessed every 3 months for patients within 2 years of registration, then every 6 months for patients in year 3
Population: eligible and treated patients
Measure: Number (80% Confidence Interval); unit: proportion of participants
Arm/Group | Arm I (Closed to Accrual as of 11/3/2008) | Arm II (Open to Accrual on 8/18/2009)
Number analyzed (Participants) | 27 | 34
proportion of participants | 0.259 [0.150 to 0.397] | 0.353 [0.243 to 0.477]
Statistical Analysis 1: Comparison: Arm I (Closed to Accrual as of 11/3/2008); Null hypothesis is that the local failure rate at 3 years is no more than 35%; Test type: Superiority or Other; p = 0.218, one sample binomial test
Statistical Analysis 2: Comparison: Arm II (Open to Accrual on 8/18/2009); The null hypothesis is that the local failure rate at 3 years is no more than 35%; Test type: Superiority or Other; p = 0.592, one sample binomial test

2. Secondary Outcome: 3-year Overall Survival Rate
Description: Overall survival (OS) is defined as time from registration to death from any cause. Patients alive are censored at the last contact date. Kaplan-Meier method was used to estimate the 3-year OS rate.
Time Frame: assessed every 3 months for patients within 2 years of registration, then every 6 months for patients in year 3
Population: eligible and treated patients
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Arm I (Closed to Accrual as of 11/3/2008) | Arm II (Open to Accrual on 8/18/2009)
Number analyzed (Participants) | 27 | 34
proportion of participants | 0.887 [0.690 to 0.962] | 0.789 [0.606 to 0.893]

3. Secondary Outcome: 3-year Progression-free Survival Rate
Description: Progression-free survival (PFS) was defined as time from registration to disease progression, relapse or death (whichever occurred first), censoring cases without PFS events at the date of last disease assessment documenting the patient was free of progression/relapse. Progression was defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions. Kaplan-Meier method was used to estimate the 3-year PFS rate.
Time Frame: assessed every 3 months for patients within 2 years of registration, then every 6 months for patients in year 3
Population: eligible and treated patients
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Arm I (Closed to Accrual as of 11/3/2008) | Arm II (Open to Accrual on 8/18/2009)
Number analyzed (Participants) | 27 | 34
proportion of participants | 0.809 [0.600 to 0.916] | 0.616 [0.432 to 0.756]

4. Secondary Outcome: Objective Response Rate
Description: Objective response rate is defined as number of patients with complete response (CR) or partial response (PR) divided by all eligible and treated patients. Responses are evaluated using the revised Response Evaluation Criteria in Solid Tumors (RECIST) guideline. CR is defined as disappearance of all target and non-target lesions. PR is defined as at least a 30% decrease in the sum of the diameters of target lesions (taking as reference the baseline sum diameters), and/or persistence of one or more non-target lesion(s).
Time Frame: Tumor assessments were made at baseline, within 4 weeks of the completion of protocol treatment, then every 6 months if patient was 1-4 years from registration, yearly if patient was 5-10 years from registration until progression/relapse using the RECIST
Population: eligible and treated patients
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Arm I (Closed to Accrual as of 11/3/2008) | Arm II (Open to Accrual on 8/18/2009)
Number analyzed (Participants) | 27 | 34
proportion of participants | 0.630 [0.424 to 0.806] | 0.647 [0.465 to 0.802]

5. Secondary Outcome: 3-year Colostomy-free Survival Rate
Description: Colostomy-free survival was defined as time from registration until time of colostomy or death without colostomy, censoring cases without colostomy at the data of last disease assessment documenting the patient was free of colostomy. Kaplan-Meier method was used to estimate the 3-year colostomy-free survival rate.
Time Frame: assessed every 3 months for patients within 2 years of registration, then every 6 months for patients in year 3
Population: eligible and treated patients who did not have permanent colostomy at study entry
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Arm I (Closed to Accrual as of 11/3/2008) | Arm II (Open to Accrual on 8/18/2009)
Number analyzed (Participants) | 27 | 34
proportion of participants | 0.849 [0.645 to 0.940] | 0.657 [0.446 to 0.804]

ADVERSE EVENTS:
Time Frame: Adverse events were assessed every cycle (1 cycle=28 days) while on treatment and for 30 days after the end of treatment. After discontinuation of treatment, severe (Grade ≥ 3) long term toxicity that had not been previously reported were collected via the Long term follow-up form using the following schedule: every 3 months within 2 years of registration, then every 6 months in years 2-5, annually afterward until year 10.
Arm/Group | Arm I (Closed to Accrual as of 11/3/2008) | Arm II (Open to Accrual on 8/18/2009)
Serious Adverse Events (participants affected / at risk) | 26/28 | 29/34
Other Adverse Events (participants affected / at risk) | 28/28 | 34/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (Closed to Accrual as of 11/3/2008) (N=28) | Arm II (Open to Accrual on 8/18/2009) (N=34)
Allergic reaction (Immune system disorders) | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 1 | 0
Anemia (Blood and lymphatic system disorders) | 2 | 5
Leukocytes decreased (Investigations) | 7 | 14
Lymphopenia (Investigations) | 3 | 6
Neutrophils decreased (Investigations) | 6 | 17
Platelets decreased (Investigations) | 2 | 4
Left ventricular systolic dysfunction (Cardiac disorders) | 0 | 1
Fatigue (General disorders) | 6 | 7
Weight loss (Investigations) | 1 | 1
INR increased (Investigations) | 1 | 0
Activated partial thromboplastin time prolonged (Investigations) | 1 | 0
Rash/desquamation (Skin and subcutaneous tissue disorders) | 0 | 1
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 0 | 2
Chemoradiation dermatitis (Injury, poisoning and procedural complications) | 4 | 0
Radiation dermatitis (Injury, poisoning and procedural complications) | 3 | 1
Ulceration (Skin and subcutaneous tissue disorders) | 1 | 1
Anorexia (Metabolism and nutrition disorders) | 3 | 7
Dehydration (Metabolism and nutrition disorders) | 9 | 11
Diarrhea w/o prior colostomy (Gastrointestinal disorders) | 15 | 23
Dry mouth (Gastrointestinal disorders) | 1 | 0
Malabsorption (Gastrointestinal disorders) | 1 | 0
Muco/stomatitis by exam, oral cavity (Gastrointestinal disorders) | 1 | 3
Muco/stomatitis (symptom) esophagus (Gastrointestinal disorders) | 0 | 1
Muco/stomatitis (symptom) oral cavity (Gastrointestinal disorders) | 2 | 1
Muco/stomatitis (symptom) pharynx (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Muco/stomatitis (symptom) rectum (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 7 | 11
Vomiting (Gastrointestinal disorders) | 2 | 5
Rectum, hemorrhage (Gastrointestinal disorders) | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1
Infection w/ gr3-4 neut, lung (Infections and infestations) | 0 | 1
Infection Gr0-2 neut, bladder (Infections and infestations) | 1 | 2
Infection Gr0-2 neut, rectum (Infections and infestations) | 1 | 0
Infection Gr0-2 neut, blood (Infections and infestations) | 0 | 1
Infection w/ unk ANC blood (Infections and infestations) | 1 | 1
Acidosis (Metabolism and nutrition disorders) | 1 | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 | 3
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 2
Creatinine increased (Investigations) | 0 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 2 | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 1 | 3
Hypokalemia (Metabolism and nutrition disorders) | 4 | 8
Hyponatremia (Metabolism and nutrition disorders) | 0 | 2
Nonneuropathic generalized weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Ataxia (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0
Abdomen, pain (Gastrointestinal disorders) | 1 | 3
Anus, pain (Gastrointestinal disorders) | 1 | 2
Back, pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Bladder, pain (Renal and urinary disorders) | 0 | 1
Head/headache (Nervous system disorders) | 1 | 1
Rectum, pain (Gastrointestinal disorders) | 2 | 1
Scrotum, pain (Reproductive system and breast disorders) | 0 | 1
Skin, pain (Skin and subcutaneous tissue disorders) | 2 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary/Upper Respiratory-other (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cystitis (Renal and urinary disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 1 | 1
Renal/GU-other (Renal and urinary disorders) | 0 | 1
Vaginal mucositis (Reproductive system and breast disorders) | 0 | 1
Thrombosis/thrombus/embolism (Vascular disorders) | 1 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (Closed to Accrual as of 11/3/2008) (N=28) | Arm II (Open to Accrual on 8/18/2009) (N=34)
Tinnitus (Ear and labyrinth disorders) | 3 | 1
Anemia (Blood and lymphatic system disorders) | 11 | 12
Leukocytes decreased (Investigations) | 15 | 11
Lymphopenia (Investigations) | 2 | 1
Neutrophils decreased (Investigations) | 11 | 7
Platelets decreased (Investigations) | 11 | 14
Sinus tachycardia (Cardiac disorders) | 0 | 2
Hypertension (Vascular disorders) | 0 | 3
Hypotension (Vascular disorders) | 2 | 2
Fatigue (General disorders) | 23 | 23
Fever w/o neutropenia (General disorders) | 4 | 6
Insomnia (Psychiatric disorders) | 1 | 4
Weight loss (Investigations) | 11 | 25
Burn (Injury, poisoning and procedural complications) | 4 | 5
Dry skin (Skin and subcutaneous tissue disorders) | 9 | 7
Alopecia (Skin and subcutaneous tissue disorders) | 9 | 5
Pruritus/itching (Skin and subcutaneous tissue disorders) | 3 | 2
Rash/desquamation (Skin and subcutaneous tissue disorders) | 2 | 2
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 15 | 19
Chemoradiation dermatitis (Injury, poisoning and procedural complications) | 2 | 1
Radiation dermatitis (Injury, poisoning and procedural complications) | 1 | 4
Hand-foot reaction (Skin and subcutaneous tissue disorders) | 2 | 0
Ulceration (Skin and subcutaneous tissue disorders) | 4 | 2
Anorexia (Metabolism and nutrition disorders) | 15 | 13
Constipation (Gastrointestinal disorders) | 7 | 7
Dehydration (Metabolism and nutrition disorders) | 2 | 5
Diarrhea w/o prior colostomy (Gastrointestinal disorders) | 15 | 9
Dysphagia (Gastrointestinal disorders) | 2 | 0
Dyspepsia (Gastrointestinal disorders) | 5 | 0
Muco/stomatitis by exam, oral cavity (Gastrointestinal disorders) | 12 | 9
Muco/stomatitis by exam, pharynx (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Muco/stomatitis (symptom) oral cavity (Gastrointestinal disorders) | 9 | 10
Nausea (Gastrointestinal disorders) | 23 | 19
Proctitis (Gastrointestinal disorders) | 0 | 2
Taste disturbance (Nervous system disorders) | 8 | 5
Vomiting (Gastrointestinal disorders) | 17 | 13
Rectum, hemorrhage (Gastrointestinal disorders) | 2 | 2
Edema limb (General disorders) | 2 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 4 | 9
Alkaline phosphatase increased (Investigations) | 1 | 4
Alanine aminotransferase increased (Investigations) | 1 | 2
Aspartate aminotransferase increased (Investigations) | 1 | 2
Hypocalcemia (Metabolism and nutrition disorders) | 4 | 8
Creatinine increased (Investigations) | 4 | 3
Hyperglycemia (Metabolism and nutrition disorders) | 2 | 3
Hypomagnesemia (Metabolism and nutrition disorders) | 17 | 21
Hypokalemia (Metabolism and nutrition disorders) | 4 | 5
Hyponatremia (Metabolism and nutrition disorders) | 3 | 7
Nonneuropathic generalized weakness (Musculoskeletal and connective tissue disorders) | 1 | 2
Dizziness (Nervous system disorders) | 3 | 1
Anxiety (Psychiatric disorders) | 0 | 2
Neuropathy-sensory (Nervous system disorders) | 5 | 3
Vision-blurred (Eye disorders) | 2 | 0
Tearing (Eye disorders) | 2 | 0
Abdomen, pain (Gastrointestinal disorders) | 3 | 4
Anus, pain (Gastrointestinal disorders) | 1 | 2
Head/headache (Nervous system disorders) | 7 | 2
Rectum, pain (Gastrointestinal disorders) | 7 | 4
Urethra, pain (Renal and urinary disorders) | 2 | 0
Vaginitis (not due to infection) (Reproductive system and breast disorders) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less